CLINICAL TRIAL: NCT07173088
Title: Efficacy and Clinical Feasibility of the Ankle Muscle Power (AMP) Program for Return to Duty After an Ankle Fracture
Acronym: AMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brian W. Noehren (Other)
Responsible Party: Sponsor-Investigator, Brian W. Noehren, Associate Dean, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103812; HT9425-25-1-0625 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-09-02; First posted 2025-09-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Ankle Fractures
Keywords: Physical Therapy; Rehabilitation
MeSH Terms: conditions — Ankle Fractures | interventions — Adenosine Monophosphate; Physical Therapy Modalities; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ankle Muscle Power (AMP) program + standard of care (Experimental): Participants will receive standard of care rehabilitation as needed and directed by the treating physical therapist. Participants will have additional exercises included to facilitate the development of power that will progress as participants move through the rehabilitation program.
  The intervention may begin approximately 12 weeks post op ± 2 weeks following fixation surgery and will have visits for up to 12 weeks with an average of 3 visits per week.
  Interventions: Other: Ankle Muscle Power (AMP) program; Behavioral: Standard of Care
- Standard of care only (Active Comparator): Standard of care rehabilitation includes range of motion, foundational strength exercises, and other modalities (i.e., icing and or low grade NMES) as needed and directed by the treating physical therapist.
  The intervention may begin approximately 12 weeks post op ± 2 weeks following fixation surgery and rehabilitation will take place for up to 12 weeks with visits occurring 3 times per week on average.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Other: Ankle Muscle Power (AMP) program — The AMP program targets various aspects of muscle power development through a program that takes the participant through 3 different stages of training over the course of their rehabilitation. This portion of the program is in addition to receiving standard rehabilitation exercises as well.
  Other Names: Physical Therapy
  Arms: Ankle Muscle Power (AMP) program + standard of care
Behavioral: Standard of Care — Standard rehabilitation program

SUMMARY:
The goal of this clinical trial is to compare two different standardized physical therapy rehabilitation programs on outcomes after an ankle fracture. Researchers will evaluate to see if the addition of ankle muscle power exercises (AMP) improve program adherence, muscle function, physical performance, and patient reported outcomes. The main questions it aims to answer are:

1. Assess feasibility and define the initial effects of the AMP program on ankle plantar flexor rate of torque development and ankle power.

   Primary hypothesis: an ankle muscle power program will have acceptable feasibility through assessment of 80% adherence, 90% treatment fidelity, recruitment (48 participants who complete the study), 80% retention, and 80% acceptability of the AMP program to facilitate clinical translation and the ability to scale-up the treatment. In addition ankle plantar flexor muscle power, plantar flexor RTD assessed isometrically, and ankle joint power, evaluated during gait and stair ascent/descent, will have significantly greater improvements in the AMP group than the standard of care group at the end of the intervention.
2. Test the effect of the AMP program on physical performance. Primary hypothesis: those completing the AMP program will have greater improvements in the 40 meter fast paced walk test and 11-stair climb test than those completing standard of care at the completion of the intervention.
3. Assess the preliminary efficacy of the AMP program on patient reported outcomes and quality of life.

Primary hypothesis: compared to standard of care, the AMP program will result in improved quality of life on the ankle fracture outcome rehabilitation measure (A-FORM)

Participants will complete rehabilitation and be assessed for outcomes at baseline and after completing the intervention. Additionally exploratory outcomes will be assessed 3 months after completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old
* Acute orthopedic injury to the ankle requiring surgical fixation
* Must have stable address and phone number to schedule follow up contact visits
* English speaking
* BMI ≤ 35 kg/m2

Exclusion Criteria:

* History of chronic pain defined as pain lasting more than 3 months and bothersome at least half the days over the past 6 months that started before the fracture
* Moderate or severe traumatic brain injury
* Initial treatment requiring amputation
* Spinal cord injury
* Unable to speak or read English
* History of schizophrenia, dementia, neurologic disorder with peripheral dysfunction, or other psychotic disorder based upon medical record or patient self-report
* Any chronic conditions that would limit their ability to participate in an intervention
* Multiple trauma that prevents engaging in intervention
* Pregnant
* Unable to participate in or complete in-person follow up visits or therapy sessions
* In Physical Therapy at the start of the intervention.
* Use of an assistive device to walk for community ambulation
* Prior lower extremity fracture within the past 2 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Adhering to the Intervention | From baseline assessment to completion of the 10 week intervention.
  Adherence refers to the commitment of a participant to participate in the rehab. Adherence will be measured by calculating the number of rehab sessions attended divided by the number of rehab sessions possible.
Percentage of Treatment That is Able to be Delivered (Fidelity) | From baseline assessment to completion of the 10 week intervention.
  Fidelity refers to the ability to perform the protocol as intended and that the participants receive the intended treatment as designed. It will be calculated as the number of deviations from protocol divided by the number of treatment sessions.
Percentage of Participants Completing the Intervention (Retention) | From baseline assessment to completion of the 10 week intervention.
  This will be calculated as the number of participants completing each intervention divided by the number of participants who start each intervention.
Percentage of Participants Who Find the Program Acceptable/Satisfactory | From baseline assessment to completion of the 10 week intervention.
  A participant satisfaction survey will be utilized to evaluate each rehabilitation protocol, care given, and rehab facility procedures. Scores will range from 1 to 5 with 1 indicating poor performance of the facility and care received versus 5 indicating excellent performance of the facility and care received.
Change in Isometric Ankle Plantar Flexor Muscle Power | Baseline assessment and post intervention visit (10-12 weeks following baseline)
  Will be assessed isotonically on a dynamometer as the change in peak power from baseline to post-intervention follow-up
Change in Ankle Rate of Torque Development (Ankle RTD) | Baseline assessment and post intervention visit (10-12 weeks following baseline)
  Will be assessed isometrically on a dynamometer as the change between baseline and post-intervention follow-up. Ankle RTD is calculated as the initial slope of the generated force curve, measured in Newton meters per second.
Change in Ankle Joint Power During Gait | Baseline and post intervention (10-12 weeks following baseline)
  Ankle joint power measured with 3D motion capture during walking
Change in Ankle Joint Power During Stairs (step up and down) | Baseline and post intervention (10-12 weeks following baseline)
  Ankle joint power measured with 3D motion capture while climbing stairs

SECONDARY OUTCOMES:
Change in Usual Gait Speed | Baseline and post intervention (10-12 weeks following baseline)
  Participants will walk at a pace that feels normal for the participant with the time to complete 5 meters recorded.
Change in Fastest Gait Speed | Baseline and following completion of the intervention (10-12 weeks post baseline visit)
  Participants will walk at their fastest comfortable speed with the time to complete 5 meters recored.
Change in 11 Stair Climb Test Score | Baseline visit and post intervention visit (10-12 weeks post baseline)
  The stair test is a measurement of functional strength, balance, and agility achieved by ascending and descending a specific number of steps (11). Scoring involves recording the total time taken to ascend and descend the steps to the nearest 100th of a second. Lower values indicate better performance.
Change in Ankle fracture outcome rehabilitation measure (A-FORM) | Baseline and post intervention (10-12 weeks following baseline)
  The Ankle Fracture Outcome of Rehabilitation Measure (A-FORM) is a patient-reported outcome measure designed to assess recovery after an ankle fracture. It focuses on physical, social, and psychological aspects of recovery. A summary score (ranging from 0 to 100) is calculated, with lower scores indicating better outcomes.
Change in PROMIS Physical Function Computer Adaptive Test | Baseline assessment and post intervention visit (10-12 weeks later)
  The PROMIS Physical Function computer adaptive test will be administered to each subject. Scale 0-100, where higher numbers indicate better physical functioning. A score of 50 is consistent with the mean score of the U.S. general population.

OTHER OUTCOMES:
Change in Brief Pain Inventory (BPI) | Baseline, following the intervention (10-12 weeks post intervention), and at a 3 month follow up after completing the intervention.
  This patient reported outcome measures assesses pain severity and interference. Scores range from 0-10 for each subscale of pain/severity or interference/impact with higher scores indicating greater pain severity and impact of pain. Scores can be compared to norms to determine if pain is considered significant.
Change in Tampa Scale of Kinesiophobia (TSK) | Baseline, following the intervention (10-12 weeks post intervention), and at a 3 month follow up after completing the intervention.
  A patient reported outcome measures that assesses fear of movement due to pain. The full TSK (17-item) yields a total score between 17 and 68, where higher scores indicate greater kinesiophobia.
Ankle Plantar Flexor muscle cross sectional area | Baseline and post intervention (10-12 weeks following the baseline visit)
  The cross sectional area of the gastrocnemius muscle will be evaluated using ultrasound imaging. The area of the muscle will be measured in cm squared.
Change in the Work Productivity and Activity Impairment Questionnaire (WPAI) | Baseline, following the intervention (10-12 weeks post intervention) and at a 3 month follow up after completing the intervention.
  A patient reported outcome measures that assesses impairments in work productivity following an injury. The WPAI questionnaire yields four scores; absenteeism, presenteeism, overall work impairment, and activity impairment which are expressed as percentages. Absenteeism is calculated as hours missed divided by total hours available for work. Presenteeism is derived from the 0-10 scale measuring health's impact on productivity while working. Overall work impairment combines both, and activity impairment measures health's effect on non-work tasks. Higher percentage scores indicate greater impairment and reduced productivity.
Change in Ankle fracture outcome rehabilitation measure (A-FORM)-midpoint | After completing isometric phase (16 ± 2 weeks post-op) and concentric phase (20 ± 2 weeks post-op)
  A summary score (ranging from 0 to 100) is calculated, with lower scores indicating better outcomes. The Ankle Fracture Outcome of Rehabilitation Measure (A-FORM) is a patient-reported outcome measure designed to assess recovery after an ankle fracture. It focuses on physical, social, and psychological aspects of recovery.
Change in Fastest Gait Speed-midpoint | After completing isometric phase (16 ± 2 weeks post-op) and concentric phase (20 ± 2 weeks post-op)
  Participants will walk at their fastest comfortable speed with the time to complete 5 meters recorded.
Change in Usual Gait Speed-midpoint | After completing isometric phase (16 ± 2 weeks post-op) and concentric phase (20 ± 2 weeks post-op)
  Participants will walk at a pace that feels normal for the participant with the time to complete 5 meters recorded.
Change in 11 Stair Climb Test Score-midpoint | After completing isometric phase (16 ± 2 weeks post-op) and concentric phase (20 ± 2 weeks post-op)
  The stair test is a measurement of functional strength, balance, and agility achieved by ascending and descending a specific number of steps. Scoring involves recording the total time taken to ascend and descend the steps to the nearest 100th of a second. Lower values indicate better performance.
Change in Isometric Ankle Plantar Flexor Muscle Power- mid point | After completing isometric phase (16 ± 2 weeks post-op) and concentric phase (20 ± 2 weeks post-op)
  Will be assessed isotonically on a dynamometer as the peak power.
Change in Ankle Rate of Torque Development (Ankle RTD)-midpoint | After completing isometric phase (16 ± 2 weeks post-op) and concentric phase (20 ± 2 weeks post-op)
  Will be assessed isometrically on a dynamometer as the slope of the generated force curve. It is the peak rate of force development measured in Newton meters per second.
Change in Ankle Hindfoot Scale (AOFAS) | Baseline assessment and post intervention visit (10-12 weeks following baseline)
  The AOFAS Ankle-Hindfoot Scale is a short survey and exam that looks at ankle and foot problems. It measures three main things: pain, how well a person can move and do daily activities, and how well the ankle and foot are lined up. The score goes from 0 to 100, with higher scores meaning less pain and better function. It helps doctors and researchers track recovery and compare treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
The dissemination plan emphasizes transparency of the study, and as a study team, the investigators are committed to sharing de-identified data for external researchers.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be available at the time of manuscript acceptance and publishing. A published manuscript is planned for mid 2029.
Access Criteria: Any external researcher will be able to access de-identified, non-PHI, individual participant data as part of the journal's supplementary information.